CLINICAL TRIAL: NCT04675554
Title: The Role of Psychological Factors and the Acceptability of New Technology in Engaging Seniors in Physical Activity: A Pilot Study
Brief Title: Role of Psychological Factors and Acceptability of New Technology in Engaging Seniors in Physical Activity
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: Laboratoire Motricité Humaine, Expertise, Sport, Santé (LAMHESS) (Unknown); Côte d'Azur Université (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20-PP-23
Record Dates: First submitted 2020-12-09; First posted 2020-12-19 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Motivation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Follow up of physical activity — participants will fill in the non-opposition form via the application and will complete, with their smartphone, a series of psychometric questionnaires. Participants will then use the mobile application for a period of 12 weeks during which time, physical activity data provided from participants smartphone will be gathered After 12 weeks, participants will complete again the same series of psychometric questionnaires.

SUMMARY:
This study will be a non-interventional study intended to identify psychological antecedents of the acceptability of WeWard application among people aged 55 years and older, , and its impacts on engagement in physical activity. Participants will be included in the study on a voluntary basis and healthy volunteers will be registered on the national volunteer database. This study will include people aged over 55 from senior citizens associations, from patients coming for frailty consultations at the Cimiez University Hospital Centre, and from any senior living in France. Regarding the recruitment, application users will receive a request to participate in a scientific study. If the request is accepted, participants will fill in the non-opposition form via the application and will complete, with their smartphone, a series of psychometric questionnaires (e.g. level of physical activity, personality, motivation, perceived physical competence, new technologies acceptability, etc.). Participants will then use the mobile application for a period of 12 weeks during which time, physical activity data provided from participants smartphone will be gathered such as the number of steps or gait speed. Psychometric questionnaires comprising each time one item (i.e. ecological momentary assessment) will be administered to participants randomly, in order to assess their evolution. After the 12 weeks of using the mobile application, older people will answer to the same series of psychometric questionnaires administered at the beginning of the study. Finally,lparticipants who will drop out the trial during this study will be contacted in order to clarify the reasons for their withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* signed non opposition
* > or = 55 years old

Exclusion Criteria:

-

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all person using the application
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
number of steps from a mobile application : | during 12 weeks
  number of steps
walking speed from a mobile application | during 12 weeks
  walking speed
walking distance from a mobile application | during 12 weeks
  walking distance
change of level from a mobile application | during 12 weeks
  change of level
Big Five Inventory | before and after 12 weeks of using the application.
  Big Five Inventory: score 1 to 5 when agree, item score is 5 when disagree, item score is 1
Perceived physical self worth | before and after 12 weeks of using the application.
  Perceived physical self worth: one item score : very bad to very good

CONTACTS AND LOCATIONS:
Overall Officials: Olivier GUERIN, PU-PH, Principal Investigator — Centre Hospitalier Universitaire de Nice

IPD SHARING:
Plan to Share IPD: Undecided